CLINICAL TRIAL: NCT05134298
Title: First Dose Pharmacokinetics for Piperacillin and Meropenem in ICU Patients
Brief Title: Pharmacokinetics of Piperacillin and Meropenem in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Petersson, Senior ICU consultant, Associate Professor, Karolinska University Hospital
Other Study IDs: K 2018-6443
Record Dates: First submitted 2019-10-28; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Antibiotic Pharmacokinetics
MeSH Terms: interventions — Piperacillin; Tazobactam; Meropenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Kohort: As specified by study population, inclusion and exclusion criteria
  Interventions: Drug: Piperacillin/tazobactam, Meropenem

INTERVENTIONS:
Drug: Piperacillin/tazobactam, Meropenem — This is an observational study exploring the antibiotic plasma concentration profiles in ICU paitents after the first drug administration.

SUMMARY:
The purpose of the study is to characterize the pharmacokinetics of meropenem and piperacillin in ICU-patients at the time of the first dose administration and to contrast that with the same measurements obtained in the same patient 2-3 days later during the course of ICU treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patient being treated in one of the participating ICUs and planned to recieve treatment with meropenem or piperacillin.

Exclusion Criteria (fullfilling any exlusion criteria means that patient cannot be included in the study):

* Not possible to retrospectively ask the patient or next of kin for consent to take part in the study or patient or next-of-kin not providing consent.
* Not posisble to obtain and process blood samples as specified by protocol.
* Ongoing renal replacement therapy.
* Patient having received the same antibiotic within the previous 96 h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU-patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume of distribution | For the first antibiotic administration and if possible for a second administration 48-72 hour later.
  Apparent volume of distribution calculated from repeated plasma concentrations measurements and pharmacokinetic modelling.
Plasma clearance | For the first antibiotic administration and if possible for a second administration 48-72 hour later.
  Plasma clearance calculated from repeated plasma concentrations measurements and pharmacokinetic modelling.

SECONDARY OUTCOMES:
Plasma antibiotic concentrations at mid and end of dosing interval | For the first antibiotic administration and if possible for a second administration 48-72 hour later.
  Plasma antibiotic concentrations at mid and end of dosing interval

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided